CLINICAL TRIAL: NCT01354925
Title: Management of Type-2 Diabetic Patients Treated With Insulin During the Ramadan An Interventional, Community Based, Comparative Study
Brief Title: Management of Type-2 Diabetic Patients Treated With Insulin During the Ramadan
Acronym: DMR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MeirMc062/2011
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Type 2; Treatment During Ramadan
Keywords: Diabetes type 2; Fasting; Ramadan; Insulin analogues
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fasting | interventions — Standard of Care

ARMS (2):
- Insulin treatment during Ramadan (Active Comparator): Insulin analogs will be used: Levemir and NovoMix70. .
  Interventions: Drug: Insulin treatment during Ramadan
- Standard treatment during Ramadan (Active Comparator): Standard of care according to physicians choice
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Insulin treatment during Ramadan — Insulin analogs will be used: Levemir and NovoMix70. The daily insulin dose will be calculated as follows: Sixty percent of the total daily dose will be used as the beginning daily dose at the first day of fasting. Sixty percent of the daily dose will be given as NovoMix70 before the Eftar (the main meal in the evening that breaks the fast). Forty percent of the amount will be given as Levemir (Early in the morning before the beginning of fasting.
  Arms: Insulin treatment during Ramadan
Drug: Standard of care — Standard of care during Ramadan according to physicians decision
  Arms: Standard treatment during Ramadan

SUMMARY:
Fasting during the Ramadan is one of the five pillars of Islam and is a mandatory duty for all healthy adult Muslims. Fasting is considered safe in young healthy subjects but it can induce harmful effects and complications in patients with diabetes. Several studies have demonstrated that patients with type 2 diabetes are prone to hypo and hyper glycemia during fasting. When treating diabetic patients with a treatment guideline the rate of these complications can be reduced. Little data is available on patients with type 2 diabetes treated with insulin. The investigators therefore propose to assess the effect of a protocol containing detemir (levemir) and a premix of insulin aspart (NovoMix70) on glucose control in patients with type 2 diabetes during the Ramadan and to compare this regimen to the standard care patients receive during this period. The investigators assume that patients receiving the intervention will have better glucose control during the Ramadan compared to patients receiving the standard care. As approximately 45 million Muslims suffer from type 2 diabetes and most of them fast during the Ramadan the results of this intervention may be significant and may improve the care of these patients allowing Muslims to respect their religious obligations without compromising their health.

ELIGIBILITY:
Inclusion Criteria:

All of these criteria should be present.

1. Patients with a diagnosis of type 2 diabetes treated with insulin (premix preparations or basal and rapid acting insulin) with or without metformin and/or a sulfonylurea drug for at least three months
2. HbA1c in the past three months ≤ 10%
3. Being capable, and willing, to perform self blood glucose monitoring and use a patient diary as required
4. Age > 18 years

Exclusion Criteria:

Any of the following:

1. Patients with a diagnosis of type 1 diabetes
2. Hypoglycemia unawareness
3. Hypersensitivity to levemir
4. Hypersensitivity to NovoMix70
5. Creatinine > 2.5 mg/l
6. AST and or ALT > 1.5 times the upper limit
7. Pregnancy
8. Mental incapacity, unwillingness or language barrier precluding adequate understanding of the study protocol or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Difference in mean 4-point SMBG during days 23-30 of treatment between the two groups. | days 23-30 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Naim Shehadeh, MD, Principal Investigator — Clalit HMO
Locations (1):
- Clalit HMO, Haifa, Israel

REFERENCES:
- [Derived] Shehadeh N, Maor Y; Ramadan Study Group. Effect of a new insulin treatment regimen on glycaemic control and quality of life of Muslim patients with type 2 diabetes mellitus during Ramadan fast - an open label, controlled, multicentre, cluster randomised study. Int J Clin Pract. 2015 Nov;69(11):1281-8. doi: 10.1111/ijcp.12695. Epub 2015 Jul 31. PMID 26234442